CLINICAL TRIAL: NCT02449642
Title: LH Hormone Pulsation in the Luteal Phase in GnRH Antagonist IVF Cycles Triggered by GnRH Agonist for Final Oocyte Maturation
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, SAMER TANNUS MD, M.D, Rambam Health Care Campus
Other Study IDs: protocol1
Record Dates: First submitted 2015-05-16; First posted 2015-05-20 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Infertility
Keywords: luteinizing hormone pulsatility; estradiol level; progesterone level
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — frequent blood tests for luteinizing hormone, estradil and progesterone levels
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- group 1: group 1 include 10 women in which blood tests will be taken on the day of oocyte pick up
- group 2: group 2 include 10 women in which blood tests will be taken on the day of embryo transfer

SUMMARY:
Monitoring the LH pulsatility during the Luteal phase in GnRH antagonist IVF cycles triggered by GnRH agonist for final oocyte maturation.

DETAILED DESCRIPTION:
About two decades ago the GnRH antagonist has been used in IVF cycles to prevent premature LH surge. In recent review GNRH antagonist has been found comparable to GnRH agonist in term of live birth rate but with reduced risk of OHSS. another advantage of using GnRH antagonist is the ability to use GnRH agonist for final oocyte maturation which has been shown to nearly eliminate the risk of OHSS. The exact mechanism of this risk reduction is still unknown.

Our aim is to do a frequent blood tests every 20 minutes for 6 hours duration in the day of ovum pick up or the day of embryo transfer to measure the level of LH, estradiol and progesterone in women triggered with GnRH agonist for final oocyte maturation.

ELIGIBILITY:
Inclusion Criteria:

* age: 18-42 years old BMI < 32 kg/m2

Exclusion Criteria:

* Hypogonadotropic hypogonadism

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women aged 18-42 years old BMI < 32 kg/M2
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
luteinizing hormone pulsatility frequency | 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam medical center, IVF unit, Haifa, Israel, Israel